CLINICAL TRIAL: NCT07254741
Title: Role of Clinical Pharmacy and Mobile Medical Applications in Detection and Minimization of Different Medication Errors in Hospitalized Patients From Adults and Children
Brief Title: Pharmacist Mobile App Intervention in Pediatric Inpatient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Abd Elhamid Mohammed Tony, Clinical Pharmacist and Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (FMBSUREC/03102023/Tony)
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Medication Safety in Pediatric Inpatients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-Led Medication Review (Experimental)
  Interventions: Behavioral: Pharmacist-Led Medication Review
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Pharmacist-Led Medication Review — Daily medication review conducted by a clinical pharmacist using mobile medical applications to identify potential medication-related problems and support safer prescribing decisions for hospitalized pediatric patients.
  Arms: Pharmacist-Led Medication Review

SUMMARY:
The goal of this study is to learn whether a clinical pharmacist-led medication review, supported by medical mobile applications, can improve the safety and quality of care for hospitalized children. The study compares usual care with enhanced pharmacist involvement to understand whether this approach reduces medication-related problems and supports better clinical outcomes.

The main questions this study aims to answer are:

Does the pharmacist-led review help identify and prevent medication issues in pediatric inpatients?

Can this intervention improve the overall quality of care during hospitalization?

Does the use of mobile medical applications assist pharmacists in making safer medication decisions?

Participants will:

Receive either routine care or routine care plus daily medication review by a clinical pharmacist

Have their medications assessed regularly to identify potential problems

Be followed during their hospital stay to observe clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

Age between 2 and 15 years

Admitted to the pediatric general inpatient ward

Prescribed three or more medications during the hospital stay

Exclusion Criteria:

Length of hospital stay less than 48 hours

Admission to the pediatric intensive care unit (PICU)

Estimated life expectancy less than 24 hours

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Medication Errors Identified | From admission to hospital discharge (an average of 3-7 days)
  Number of medication errors detected during routine review of inpatient medication orders, including prescribing, dosing, frequency, and administration-related issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Coordination Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No